CLINICAL TRIAL: NCT01052922
Title: Systems of Support (SOS) to Increase Colon Cancer Screening and Follow-up Supplement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Fred Hutchinson Cancer Center (Other); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 3R01CA121125-03S1 (NIH)
Record Dates: First submitted 2010-01-19; First posted 2010-01-21 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Colorectal Cancer Screening
Keywords: Colorectal Neoplasms; Mass Screening; Population Surveillance; Randomized controlled trial; Occult Blood; Colonoscopy; Sigmoidoscopy; Health Behavior
MeSH Terms: conditions — Colorectal Neoplasms; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 2 sample InSure (Active Comparator)
  Interventions: Other: 2 sample InSure
- 1 sample OC-Micron (Active Comparator)
  Interventions: Other: 1 sample OC-Micron
- 3 sample g-SENSA (Active Comparator)
  Interventions: Other: 3 sample g-SENSA

INTERVENTIONS:
Other: 3 sample g-SENSA — Participants will be mailed to a 3 sample g-SENSA FOBT kit to complete at home and mail back to the lab for screening.
  Arms: 3 sample g-SENSA
Other: 2 sample InSure — Participants will be mailed to a 2 sample InSure FOBT kit to complete at home and mail back to the lab for screening.
  Arms: 2 sample InSure
Other: 1 sample OC-Micron — Participants will be mailed to a 1 sample OC-MICRON FOBT kit to complete at home and mail back to the lab for screening.
  Arms: 1 sample OC-Micron

SUMMARY:
Ancillary Aim #1 We will evaluate intervention effects by comparing binary outcomes for screening (yes/no) in the primary SOS study. In this aim, we propose to calculate actual screening rates by use of time-to-event analyses (also known as survival analysis). The outcome variable of interest is the first time since randomization to have CRCS, either based on FOBT, FS, or CS. Knowing screening rates will not only enable us to make comparisons between groups, but also over time.

Ancillary Aims #2 and #3 We will recruit additional participants for two ancillary study aims. First, we will enroll patients age 50-74 years using the same criteria as for the primary SOS study, which includes neither history of colorectal cancer nor evidence of life-limiting disease. Participants who return the questionnaire, consent and considered eligible will be randomized to receive one of three different at-home fecal test kits. The kits will be returned to the GH centralized laboratory, and participants will be informed about lab results using standard GH pathways. Participants who have a test-positive will receive a series of two follow-up surveys (first at 1-2 weeks post result and second at 4-months post result). A comparison group of test-negative results will be matched based on selected criteria, and this group will also receive the follow-up surveys. Participants at both time intervals who do not return the survey via mail will be called and if available, administered the questionnaire via phone.

ELIGIBILITY:
Inclusion Criteria:

* Not up to date on CRCS
* Continuously enrolled in GHC for 24 months
* Expected to continue to be enrolled at GHC for 24 months

Exclusion Criteria:

* Known high risk for CRC
* History of CRC
* History of inflammatory bowel disease
* Current anticoagulation therapy
* Organ failure
* Serious illness
* Debilitating disease
* Dementia
* Nursing home resident.

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2260 (Actual)
Dates: Start 2009-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Adherence to FOBT test kit | 1-2 months

CONTACTS AND LOCATIONS:
Overall Officials: Beverly B Green, MD,MPH, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Washinton Health Research Institute, Seattle, Washington, United States

REFERENCES:
- [Derived] Chubak J, Bogart A, Fuller S, Laing SS, Green BB. Uptake and positive predictive value of fecal occult blood tests: A randomized controlled trial. Prev Med. 2013 Nov;57(5):671-8. doi: 10.1016/j.ypmed.2013.08.032. Epub 2013 Sep 9. PMID 24029556